CLINICAL TRIAL: NCT07082478
Title: External Carotid Blood Flow Dynamics in Individuals With Post-Bariatric Hypoglycemia (PBH): Pilot Study
Brief Title: External Carotid Blood Flow in Individuals With Post-Bariatric Hypoglycemia
Status: Recruiting | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Mary Elizabeth Patti, Senior Investigator, Joslin Diabetes Center
Other Study IDs: STUDY00000303
Record Dates: First submitted 2025-06-10; First posted 2025-07-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hypoglycemia; Cerebral Blood Flow
Keywords: hypoglycemia; postprandial hypoglycemia; bariatric surgery; autonomic dysfunction; cerebral blood flow
MeSH Terms: conditions — Hypoglycemia; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy individuals: individuals with no history of hypoglycemia or upper gastrointestinal surgery
  Interventions: Device: in-ear device measuring blood flow

INTERVENTIONS:
Device: in-ear device measuring blood flow — A small in-ear wearable device will be placed to monitor the blood flow to the head. The investigators will make sure it fits comfortably and show the participant how to use it properly.
  Dexcom G6 Pro: This continuous glucose monitor (CGM) will be placed under the skin of the abdomen to monitor sensor sugar levels.
  These sensors will be placed during visit one and will be worn together for 10 days. A followup visit (visit 2) will occur remotely at 4-6 days later. A final visit will occur after 10 days when the device will be removed.

SUMMARY:
This is a pilot study (small-scale study) that aims to understand more about how blood flow changes in people who have low blood sugar after bariatric surgery (post-bariatric hypoglycemia) compared to those who have had surgery without hypoglycemia, those who have hypoglycemia without surgery, or those who do not experience low blood sugar.

This study has two phases. This is the first phase, and the purpose is to test comfort and feasibility of a novel in-ear wearable device (Lumia Health) that measures blood flow changes to the head. Information from the study will help the investigators determine if the device is suitable to be used in the second phase of the study.

DETAILED DESCRIPTION:
Visit 1 (Screening) This visit will last about 2 hours. Participants will be asked to come to Joslin Diabetes Center.

During the screening visit, a study team member will go over the informed consent form with participants and will explain why this study is being done and the study procedures involved. Participants will have to sign the consent form before any study related procedures take place. After participants sign the consent, the following procedures will be done to ensure eligibility and that it is safe to be part of the study.

* Review medical history by the study doctor.
* Participants will be asked to sign a release of information form so that the investigators may obtain additional information about medical history from prior physicians and hospitals. Medical records including laboratory results (within the last 6 months) will be reviewed by the study doctor.
* Physical examination, vital signs and anthropometrics (blood pressure, heart rate, temperature, height and weight) and an otoscopic exam (a look inside the external ear).
* Urine pregnancy test (if participant is a female of child bearing potential) that must be negative in order to continue participation.
* Questionnaires: Investigators will ask participants to fill out several questionnaires that will help the investigators assess any symptoms of low blood sugar or autonomic symptoms:

  * Edinburgh Hypoglycemia Symptom Scale (EHSS)
  * Dumping Symptom Rating Scale (DSRS) questionnaire
  * Composite Autonomic Symptom Score (COMPASS 31)
  * Orthostatic Hypotension Questionnaire (OHQ)
* Devices: If the participant is eligible, a member of the study team will place the following devices. The participant will wear both devices for 10 days (24 hours per day) · Lumia Health: A small in-ear wearable device will be placed to monitor the blood flow to the head. The study team will make sure it fits comfortably and show the participant how to use it properly. A member of the Lumia team may be present during the placement of the device in order to assist the study team with choosing the best size of the device to match the shape of the participant's ear. If the participant is uncomfortable with this, study team members will be able to perform this procedure (after receiving instructions from a Lumia team member).

Procedure: (1) Removing earrings or jewelry if needed and cleaning the outer ear to ensure a secure fit. (2) Positioning the device on the frontal surface of the left ear cartilage. (3) Adjusting it to fit comfortably. If participant experiences any discomfort during placement, they will be asked to inform the study team.

Employees at Lumia Health will process signals from the device and provide the Joslin team with the blood flow information. This information will be de-identified, meaning it will not include any personally identifiable data.

Dexcom G6 Pro: This continuous glucose monitor (CGM) will be placed under the skin on the abdomen to monitor the participant's sensor glucose (sugar) levels.

Insertion Procedure: (1) A suitable location on the abdomen is identified. (2) The CGM is placed against the skin at the chosen site. The sensor is inserted in the skin with a simple press or click; this causes little to no discomfort. (3) A small transmitter is connected to the sensor to allow glucose readings to be transmitted to a monitoring device (receiver), which the participant will keep with them during the duration of the monitoring period.

Diaries: Investigators will ask participants to keep a written paper diary of daily meals, liquids (including caffeinated beverages), physical activity and any issues with the device (Lumia).

At the end of the visit, the participant will be scheduled for the next 2 visits. Additionally, the participant will be provided contact information for the study team in case any questions or issues arise during the study.

Visit 2 (Follow up)

This visit will happen remotely, between days 4-6 after Visit 1. A study team member will call the participant by video or phone. This visit will include:

Wellness check: The investigators will check how the participant is doing, see if there are any problems, and ask about experience with both the ear and CGM devices.

Ear device check: A member of the study team will review the data collected on the cloud from previous days to ensure the ear device is functioning properly. If everything is working well, the investigators will encourage participants to continue wearing the device . If there are issues with data collection or problems with device, the investigators will provide instructions to improve data collection and schedule a follow-up call if needed.

Questions and support: Investigators will be available to answer any questions that the participant may have.

At the end of this call visit, the investigators will provide instructions for the next visit.

Visit 3 (End of Study)

This visit will last approximately 2 hours at the Joslin Diabetes Center. The visit will include the following:

Review medical history, including any updates since the last visit. Physical examination, vital signs (blood pressure, heart rate, temperature, height and weight) and an otoscopic exam (a look inside the external ear).

Review of diaries the participant completed during the study. The participant will be asked to complete the same surveys as at Visit 1 and additional surveys about the experience with the device.

The participant will return study devices to the study team so the information can be downloaded for analysis.

The investigator will review the glucose monitoring information with the participant at the end of this visit, but will not be able to review data from the ear device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years of age, inclusive at screening.
* Individuals able to provide informed consent and follow all study procedures, including complete daily food, activity, and symptom diaries, and willingness to provide access to medical record review.
* For healthy control group: individuals without a history of upper gastrointestinal surgery and without reported symptoms of hypoglycemia.
* Individuals with access to personal iPhone running operating system 16 (iOS) or later versions (not feasible for Android platform users) and a password-protected home Wi-Fi network.

Exclusion Criteria:

* History of coronary artery disease or presence of 2 or more risk factors including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use.
* History of myocardial infarction, unstable angina or revascularization within the past 6 months.
* History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia.
* Documented hypoglycemia occurring in the fasting state (> 12 hours fast).
* Concurrent administration of β-blocker therapy.
* Vigorous physical activity within 24 hours prior to assessment.
* Seizure disorder (other than with suspect or documented hypoglycemia).
* Hematocrit < 33% (women) or <36% (men) within the past 6 months.
* History of insulinoma.
* Use of central nervous system-active medications, including: antidepressants, anxiolytics, antipsychotics, stimulants, antiepileptics, sedatives and opioids.
* History of severe neurologic vascular disease (e.g. cerebrovascular disease/stroke).
* History of previous diseases associated with dysautonomia (e.g. multiple system atrophy, multiple sclerosis, Parkinson's disease).
* Impaired hepatic function (aspartate amino transaminase and/or alanine amino transaminase >2x upper limit of normal range), as determined within the past 6 months.
* Impaired renal function (serum creatinine >1.5 mg/dL), as determined within the past 6 months.
* Serious psychiatric or substance abuse disorders (e.g. alcohol, opioid, cocaine use disorder), as judged by the study investigator.
* Non-consent or inability to comply with study procedures.
* Current pregnancy and/ or lactation.
* Vulnerable individuals (e.g., fetuses, children, prisoners) and those judged by the investigator to be unsuitable for the study.
* Individuals wearing earrings or other jewelry in the left ear who are unable or unwilling to remove them for the duration of the study.
* Unwillingness to wear study masked CGM for duration of study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy individuals without hypoglycemia or upper gastrointestinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of study completion | up to 10 days
  Feasibility as determined by rate of study completion
Number of days with viable data (complete recordings) | up to 10 days
  Feasibility as determined by number of days with viable data (complete recordings)
Participant-reported outcome scores | up to 10 days
  Scores from a qualitative survey (Patient-Reported Outcomes for In-Ear Device, adapted from the COPROD questionnaire (COnfort des PROtections auDitives/COmfort of hearing PROtection Devices) of patient acceptance of in-ear wearable device at study completion.
Correlation between external cerebral blood flow (eCBF) (arbitrary units) and corresponding sensor glucose values (mg/dL) | up to 10 days
  Determine correlation between external cerebral blood flow (arbitrary units) and nearest sensor glucose levels (mg/dL), summed over the length of wear for each participant
Correlation between rate of change in eCBF (arbitrary units) and rate of change in sensor glucose (mg/dL) | up to 10 days
  Determine correlation between rate of change from baseline in eCBF and rate of change in sensor glucose values, summed over the length of wear for each participant

SECONDARY OUTCOMES:
Success of data transfer from ear device to study database | up to 10 days
  Success of blood flow data transfer (yes/no) from ear device to study database for each participant
Percentage of time with successful blood flow (arbitrary units) data collection | up to 10 days
  The percentage of time with successful data collection, normalized to total wear time (hours)
Change in eCBF over 3 hours after meal initiation | up to 10 days
  Change in eCBF over 3 hours after meal initiation, as compared with mean eCBF over 1 hour prior to meal ingestion
Change in eCBF during physical activity, measured by integrated eCBF changes from onset of activity to completion of activity. | up to 10 days
  Change in eCBF from baseline during physical activity, measured by integrated eCBF changes from onset of activity to completion of activity
Correlation of hypoglycemia symptom score, measured by the Edinburgh Hypoglycemia Scale (EHHS) at study entry, with the frequency of low sensor glucose readings (% of time with sensor glucose < 70 mg/dL) | up to 10 days
  The total Edinburgh Hypoglycemia Score (obtained via survey at study entry) will be correlated with the % of time with sensor glucose readings below 70 mg/dL) for each participant
Correlation of dysautonomia symptom score, measured by the COMPASS survey at study entry, with the frequency of low sensor glucose readings (% of time with sensor glucose <70 mg/dL) | up to 10 days
  The COMPASS score will be correlated with the % of time with sensor glucose readings below 70 mg/dL for each participant.
Correlation of hypoglycemia symptom score, measured by the Edinburgh Hypoglycemia Score at study entry, with the coefficient of variation in eCBF (SD/mean) over the duration of the study | up to 10 days
  The EHSS score will be correlated with the coefficient of variation in eCBF over the duration of the study
Correlation of dysautonomia symptom score, measured by the COMPASS survey at study entry, with the coefficient of variation in eCBF (SD/mean) over the duration of the study | up to 10 days
  The COMPASS score will be correlated with the coefficient of variation in eCBF over the duration of the study.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, up to 10 days
  Adverse events will be recorded and graded for severity and relatedness by study staff during course of study

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Patti, M.D., Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared for this pilot study.

REFERENCES:
- [Background] Gold AE, MacLeod KM, Frier BM. Frequency of severe hypoglycemia in patients with type I diabetes with impaired awareness of hypoglycemia. Diabetes Care. 1994 Jul;17(7):697-703. doi: 10.2337/diacare.17.7.697. PMID 7924780
- [Background] Kaufmann H, Malamut R, Norcliffe-Kaufmann L, Rosa K, Freeman R. The Orthostatic Hypotension Questionnaire (OHQ): validation of a novel symptom assessment scale. Clin Auton Res. 2012 Apr;22(2):79-90. doi: 10.1007/s10286-011-0146-2. Epub 2011 Nov 2. PMID 22045363
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Laurenius A, Olbers T, Naslund I, Karlsson J. Dumping syndrome following gastric bypass: validation of the dumping symptom rating scale. Obes Surg. 2013 Jun;23(6):740-55. doi: 10.1007/s11695-012-0856-0. PMID 23315151
- [Background] Deary IJ, Hepburn DA, MacLeod KM, Frier BM. Partitioning the symptoms of hypoglycaemia using multi-sample confirmatory factor analysis. Diabetologia. 1993 Aug;36(8):771-7. doi: 10.1007/BF00401150. PMID 8405746
- [Background] Addison P, Carsky K, Patti ME, Roslin M. Hypoglycemia and Dysautonomia After Bariatric Surgery: a Systematic Review and Perspective. Obes Surg. 2022 May;32(5):1681-1688. doi: 10.1007/s11695-022-05960-x. Epub 2022 Feb 8. PMID 35133603
- [Background] Zhang JB, Tamboli RA, Albaugh VL, Williams DB, Kilkelly DM, Grijalva CG, Shibao CA. The incidence of orthostatic intolerance after bariatric surgery. Obes Sci Pract. 2019 Dec 6;6(1):76-83. doi: 10.1002/osp4.383. eCollection 2020 Feb. PMID 32128245
- [Background] Tripathi H, Gonuguntla A, Lee D, Fudim M, Brinker J, Tandri H. Monitoring Carotid Blood Flow Using In-Ear Wearable Device During Tilt-Table Testing. JACC Clin Electrophysiol. 2023 May;9(5):710-712. doi: 10.1016/j.jacep.2023.02.002. Epub 2023 Mar 22. No abstract available. PMID 36951817
- [Background] An Z, Wang H, Mokadem M. Role of the Autonomic Nervous System in Mechanism of Energy and Glucose Regulation Post Bariatric Surgery. Front Neurosci. 2021 Nov 23;15:770690. doi: 10.3389/fnins.2021.770690. eCollection 2021. PMID 34887725